CLINICAL TRIAL: NCT01871961
Title: Evaluation of Rheumatoid Arthritis Patient Performance Using the Metoject® Prefilled Pen (Methotrexate 50 mg/mL, Prefilled Pen) for Subcutaneous Injection and Subsequent Pharmacokinetic Assessment of Drug Delivery
Brief Title: Evaluation of Patient Performance Using the Metoject Device for Subcutaneous Injection in Rheumatoid Arthritis (RA)Patient
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: medac GmbH (Industry)
Collaborators: PPD Development, LP (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC-MTX.15/HF
Record Dates: First submitted 2013-05-14; First posted 2013-06-07 (Estimated); Last update posted 2015-03-17 (Estimated); Status verified 2015-03

CONDITIONS: Rheumatoid Arthritis (RA)
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Methotrexate

ARMS (1):
- Methotrexate (Experimental)
  Interventions: Drug: Methotrexate (Metoject® prefilled pen)

INTERVENTIONS:
Drug: Methotrexate (Metoject® prefilled pen)

SUMMARY:
To evaluate the human factors/usability of Rheumatoid Arthritis (RA) patients with the Metoject® prefilled pen (including a label comprehension assessment and a device robustness evaluation).

ELIGIBILITY:
Inclusion Criteria:

* Is a suitable candidate for treatment with Methotrexate for Rheumatoid Arthritis
* Male or female patient who is 16 years of age or older

Exclusion Criteria:

* Is a female patient who is pregnant, trying to become pregnant, or breast feeding, or of childbearing potential, sexually active and not practicing a highly reliable method of birth control during the study and at least 6 months thereafter
* Has any history of hypersensitivity to the investigational medicinal product
* Has a history of or current inflammatory arthritis or rheumatic autoimmune disease other than Rheumatoid Arthritis (RA)
* Is unable to comprehend written labeling and training materials

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2012-10; Primary Completion 2013-02 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
To evaluate the human factors/usability of Rheumatoid Arthritis (RA) patients with the Metoject® prefilled pen (including a label comprehension assessment and a device robustness evaluation). | 1 year
  Questionnaires to assess the comprehension of the label (instruction for use of the prefilled pen) and device robustness evaluation after usage of the prefilled pen

CONTACTS AND LOCATIONS:
Locations (1):
- Rheumatology Arthitis & Rheumatic Care center, South Miami, Florida, United States